CLINICAL TRIAL: NCT06500065
Title: Clinical Feasibility and Potential Clinical Benefit of 68Ga-DOTATATE PET/CT Assessment of Soft Tissue Sarcomas for Potential Peptide Receptor Radionuclide Therapy
Brief Title: 68Ga-DOTATATE PET/CT for the Diagnosis of Soft Tissue Sarcomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Gabriel Tinoco, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-20208; NCI-2020-11528 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — 68Ga-DOTA-iodo-Tyr(3)-octreotate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (68Ga-DOTATATE dPET/CT) (Experimental): Patients receive gallium Ga 68-HA-DOTA-TATE intravenously (IV) and undergo dPET/CT over 60 minutes up to two weeks after starting standard chemotherapy. Beginning 24 hours after gallium Ga 68-HA-DOTA-TATE dPET/CT, patients also receive fludeoxyglucose F-18 IV and undergo dPET/CT over 60 minutes..
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga 68-HA-DOTA-TATE; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo dPET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: Gallium Ga 68-HA-DOTA-TATE — Given IV
  Other Names: 68Ga-DOTA-3-iodo-Tyr3-octreotate; 68Ga-DOTA-iodoTyr3-octreotate; 68Ga-HA-DOTATATE; [68Ga]DOTA-3-iodo-Tyr3-octreotate; [68Ga]high-affinity DOTATATE
Procedure: Positron Emission Tomography — Undergo dPET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well 68Ga-DOTATATE digital PET/CT work in diagnosing soft tissue sarcoma. 68Ga-DOTATATE is a radiotracer that may improve image quality of PET imaging. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 68Ga-DOTATATE. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. 68Ga-DOTATATE digital PET/CT may work better in imaging patients with soft tissue sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and capability of gallium Ga 68-HA-DOTA-TATE (68Ga-DOTATATE) digital positron emission tomography (dPET)/ computed tomography (CT) imaging for soft tissue sarcomas.

SECONDARY OBJECTIVES:

I. To evaluate the clinical benefit of 68Ga-DOTATATE for a comprehensive assessment of soft tissue sarcomas (STS) using next-generation digital PET detector technology.

II. To describe the perfusion and early tumor uptake kinetics of tumor targets at baseline and following conventional systemic therapy using both 68Ga-DOT AT A TE dPET/CT and 18F-FDG dPET/CT approaches.

III. Using list-mode dPET acquisitions following standard 68Ga-DOTATATE dose administrations, imaging datasets will be retrospectively generated to simulate lower dose or faster image acquisition in order to define further the minimum 68Ga-DOTATATE dose and PET image acquisition times needed to maintain lesion detectability and PET quantification.

V. To assess the feasibility for 68Ga-DOTATATE dPET/CT to identify and stratify STS patients with SSTR2-positive soft tissue sarcoma lesions for future therapy planning using 177Lu-DOTATATE peptide receptor radionuclide therapy (PRRT) for patients with 68Ga-DOTATATE-avid sarcomas.

VI. To assess the safety of 68Ga-DOTATATE in this patient population.

OUTLINE:

Patients receive gallium Ga 68-HA-DOTA-TATE intravenously (IV) and undergo dPET/CT over 60 minutes up to two weeks after starting standard chemotherapy. Beginning 24 hours after gallium Ga 68-HA-DOTA-TATE dPET/CT, patients also receive fludeoxyglucose F-18 IV and undergo dPET/CT over 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age
* Patients diagnosed with any stage of soft tissue sarcomas candidates for systemic therapies
* Patients with one standard of care PET/CT scan up to 30 days before enrollment at the Ohio State University facilities.

Exclusion Criteria:

* Hypersensitivity to somatostatin or similar peptides
* Somatostatin long-acting analog in the past 6 months
* Patients who are pregnant or lactating
* Patients who are currently incarcerated
* Patients with acute infections
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Patients exceeding the weight limitations of the scanner or are not able to enter the bore of the dPET/CT scanner due to body mass index (BMI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Regions of pathologically increased tracer uptake | At completion of imaging
  Positron emission tomography (PET) images will be evaluated visually for regions of pathologically increased tracer uptake that could not be attributed to normal physiologic activity. The non-contrast enhanced computed tomography images are used for attenuation correction and for fusion with PET images to allow for anatomical - localization of PET findings.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 7 days after completion of imaging
  The incidence of adverse events for each patient will be reported using CTCAE v.5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel R Tinoco Suarez, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States